CLINICAL TRIAL: NCT00587314
Title: The Effect of Ablation Therapy on Barrett's Esophagus
Acronym: ablation IN BE
Status: Enrolling by invitation | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Cadman Leggett, Principal Investigator, Mayo Clinic
Other Study IDs: 258-04
Record Dates: First submitted 2007-12-21; First posted 2008-01-07 (Estimated); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Barrett's Esophagus; Early Esophageal Adenocarcinoma
Keywords: Photodynamic Therapy; Barrett's Esophagus; Early Esophageal Adenocarcinoma
MeSH Terms: conditions — Barrett Esophagus; Adenocarcinoma Of Esophagus | interventions — Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Esophageal Biopsy
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients with Barrett's Esophagus or early esophageal adenocarcinoma who will or have had ablation therapy will be enrolled in this long term follow up study
  Interventions: Other: Biopsy

INTERVENTIONS:
Other: Biopsy — Biopsies for research purposes will be obtained when returning for clinically indicated surveillance of Barrett's Esophagus

SUMMARY:
To assess the effect of ablative therapy (Photodynamic Therapy or Radiofrequency ablation ) on Barrett's Esophagus

DETAILED DESCRIPTION:
To assess the effect of ablation therapy on Barrett's esophagus. Proposal Ablation therapy is an FDA approved treatment to decrease cancer risk in Barrett's esophagus mucosa. This is being performed in our Barrett's Esophagus Unit on a regular basis. However, the longterm outcomes of this therapy is not established and there are patients who have been treated who later re-develop Barrett's mucosa. This study will allow us store tissue samples that can later be used to assess the effect of ablative therapy on Barrett's esophagus.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have had or qualify for ablation therapy for treatment of their barrett's esophagus with high grade dysplasia or early esophageal adenocarcinoma
* Ability to provide informed consent

Exclusion Criteria:

* Eastern Cooperative Oncology Group performance status 3 or 4
* Inability to tolerate endoscopic procedures
* Pregnancy: Females of child-bearing age will be screened with pregnancy test.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have had or qualify for ablation therapy for treatment of their barrett's esophagus
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2004-01; Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Response to treatment | at time of surveillance intervals
  presence of persistent or recurrence of barrett's esophagus and/or dysplasia

CONTACTS AND LOCATIONS:
Overall Officials: Cadman Leggett, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States